CLINICAL TRIAL: NCT04893993
Title: PBC Induced Fatigue Treated With Thiamine (PIFT) - The Effect of Oral Thiamine Supplement in 4 Weeks to Patients With Primary Biliary Cholangitis (PBC) and Chronic Fatigue. A Randomised Placebo Controlled Crossover Study
Brief Title: PBC Induced Fatigue Treated With Thiamine
Acronym: PIFT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henning Grønbæk (Other)
Collaborators: Aarhus University Hospital (Other); Hospitalsapoteket Region Midtjylland (Unknown); GCP-unit at Aarhus University Hospital, Aarhus, Denmark (Other); Region Hovedstadens Apotek (Other Government)
Responsible Party: Sponsor-Investigator, Henning Grønbæk, MD., Clinical professor, consultant, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PIFT AU
Record Dates: First submitted 2021-05-04; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Thiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thiamine-Placebo (Other): 12 weeks: 4 weeks with Thiamine, 4 weeks wash-out, 4 weeks placebo
  Both placebo and Thiamine are oral tablets of 300mg pr. tablet. The dosage depends on gender and weight of the participants, with a maximum of 1800mg intake pr. day.
  Interventions: Drug: Thiamine; Drug: Placebo
- Placebo-Thiamine (Other): 12 weeks: 4 weeks placebo, 4 weeks wash-out, 4 weeks with Thiamine
  Both placebo and Thiamine are oral tablets of 300mg pr. tablet. The dosage depends on gender and weight of the participants, with a maximum of 1800mg intake pr. day.
  Interventions: Drug: Thiamine; Drug: Placebo

INTERVENTIONS:
Drug: Thiamine — Tablets. 300mg/tablet. Dosage depends on gender and weight
Drug: Placebo — Tablets. Same number of tablets as Thiamine

SUMMARY:
Primary biliary cholangitis (PBC) is a chronic autoimmune liver disease characterised by destruction of the intrahepatic bile ducts leading to liver inflammation and fibrosis, and ultimately liver cirrhosis and end-stage liver disease. More than 50% of patients with PBC suffer from chronic fatigue, and approximately 20% suffer from severe fatigue with negative impact on their quality of life. Although fatigue is a large problem in patients with PBC, no effective treatments are available.

A Danish intervention study have shown that high dose oral thiamine (Vitamin B1) were effective in treating chronic fatigue in patients with inflammatory bowel disease. In this study, only few and minor adverse events to thiamine treatment were observed. Although the precise mechanism of work remains unknown, the investigators see no reason that this cannot be transferred topatients with PBC. Hence, the investigators aim to conduct a study investigating the use of oral thiamine in chronic fatigued patients with PBC.

The study will be conducted as a double-blinded, placebo-controlled, randomised, crossover trial including 36 patients with PBC and with a higher fatigue level than in the general population for more than six months. The patients will be randomised into one of two 3x4 weeks setups; 1) thiamine for four weeks followed by four weeks washout and finally four weeks of placebo or 2) placebo for four weeks followed by four weeks washout and finally four weeks of thiamine. The primary endpoint is to investigate the fatigue-level before and after treatment with thiamine and placebo using every patient as their own control. Fatigue-level will be measured using international validated questionnaires. The doses of thiamine are calculated based on the patient gender and weight. All patients will be included in the outpatient clinic at the Department of Hepatology and Gastroenterology at Aarhus University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* PBC for more than 3 months
* PBC-40 fatigue score >32
* Fatigued for at least 6 months

Exclusion Criteria:

* Comorbidity that can explain fatigue
* Non-compliant patients
* Pregnancy
* Expected surgical interventions during the study period
* Chronic kidney disease (eGFR<60)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue | After 4 weeks active treatment
  Change in levels of fatigue measured by the Primary biliary cholangitis-40 (PBC-40) fatigue domain. The fatigue domain measures the severity of fatigue on a scale from 11-55, where 55 is maximun fatigue. A change in PBC-40 fatigue domain of 5 points or more is regarded as a clinical relevant change.

SECONDARY OUTCOMES:
Disease-specific Quality of Life | Week 4, 8 and 12
  Changes in Health-related Quality of life, measured by the disease specific Primary biliary Cholangitis-40 (PBC-40).
Health-related Quality of Life | Week 4, 8 and 12
  Changes in Health-related Quality of Life, measured by the generic EQ-5D-5L tool (mainly the VAS-scale from 0-100, where 100 is best).
Fatigue | Week 8 and 12
  Change in levels of fatigue measured by the Primary biliary cholangitis-40 (PBC-40) fatigue domain. The fatigue domain measures the severity of fatigue on a scale from 11-55, where 55 is maximun fatigue. A change in PBC-40 fatigue domain of 5 points or more is regarded as a clinical relevant change.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus University Hospital, Denmark, Aarhus N, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bager P, Bossen L, Gantzel R, Gronbaek H. High-dose oral thiamine versus placebo for chronic fatigue in patients with primary biliary cholangitis: A crossover randomized clinical trial. PLoS One. 2024 Mar 29;19(3):e0301354. doi: 10.1371/journal.pone.0301354. eCollection 2024. PMID 38551983